CLINICAL TRIAL: NCT00505128
Title: Impact on Outcome of Early Endoscopic Extraction of Bile Duct Stones in Biliary Pancreatitis: a Prospective Multicenter Randomized Controlled Study
Brief Title: Impact on Outcome of Early Endoscopic Extraction of Bile Duct Stones in Biliary Pancreatitis
Acronym: EEPAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Cecile jourdain, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P051054
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2007-05

CONDITIONS: Biliary Pancreatitis
Keywords: Biliary pancreatitis; Bile duct stones; EUS Endoscopic UltraSonography; Endoscopic sphincterotomy; ERCP
MeSH Terms: conditions — Cholecystolithiasis | interventions — Sphincterotomy, Endoscopic; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): to test the interest of early bile duct decompression by endoscopic sphincterotomy after early non invasive diagnosis by endosonography or MR cholangiography
  Interventions: Procedure: Endoscopic sphincterotomy

INTERVENTIONS:
Procedure: Endoscopic sphincterotomy — procedure
  Other Names: procedure

SUMMARY:
Impact on outcome of early endoscopic extraction of bile duct stones in biliary pancreatitis: a prospective multicenter randomized controlled study.

DETAILED DESCRIPTION:
Impact on outcome of early endoscopic extraction of bile duct stones in biliary pancreatitis: a prospective multicenter randomized controlled study.

Main objective: to test the interest of early bile duct decompression by endoscopic sphincterotomy after early non invasive diagnosis by endosonography or MR cholangiography.

Prospective multicenter randomized controlled study with direct patient benefit

ELIGIBILITY:
Inclusion Criteria:

* Previous medical examination
* Age over 18
* Acute biliary pancreatitis
* Timespan between onset of symptoms and randomization <72h
* No involvement in another clinical study
* Informed consent obtained

Exclusion Criteria:

* Non biliary pancreatitis
* Age < 18
* Timespan between onset of symptoms and randomization >72h
* No follow-up possible beyond 3 months after inclusion
* Ongoing pregnancy
* No informed consent
* No health insurance affiliation
* Involvement in another clinical study
* Incapacity to understand subject information
* Counter indication of MRI examination if echo-endoscopy is not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients cured or consolidated as a function of time | during 12 months

SECONDARY OUTCOMES:
overall morbidity | during the 36 months
overall mortality | during the 36 months
endoscopic procedure-related morbidity and mortality | during the 12months
LOS | during the 12 months
morbidity in the subgroup of patients with bile duct stones left in situ (secondary sphincterotomies) | during the 12 months
economic data | during the 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederic PRAT, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Cochin, Paris, France